CLINICAL TRIAL: NCT02877082
Title: Phase II Trial of Low Toxicity GVHD Prevention and Enhanced Immune Recovery With Tacrolimus, Bortezomib and Thymoglobulin® TBT
Brief Title: Tacrolimus, Bortezomib, & Thymoglobulin in Preventing Low Toxicity GVHD in Donor Blood Stem Cell Transplant Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Zaid Al-Kadhimi, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00082499; NCI-2016-01035 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship3258-16 (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-03

CONDITIONS: Acute Leukemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Diffuse Large B-Cell Lymphoma; Follicular Lymphoma; Graft Versus Host Disease; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Graft vs Host Disease; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders | interventions — thymoglobulin; Antilymphocyte Serum; Bortezomib; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus, bortezomib, thymoglobulin (Experimental): Patients receive tacrolimus IV on day -3 through day 180. Patients may receive tacrolimus PO later at the doctor's discretion. Patients receive thymoglobulin IV on days -3, -2, and -1 and bortezomib IV on day 0 and day 3. Patients undergo allogeneic bone marrow transplant on day 0.
  Interventions: Biological: Thymoglobulin; Drug: Bortezomib; Drug: Tacrolimus

INTERVENTIONS:
Biological: Thymoglobulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Anti-Thymocyte Globulin
Drug: Bortezomib — Given IV
  Other Names: LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase II trial studies how well tacrolimus, bortezomib, and anti-thymocyte globulin (thymoglobulin) work in preventing low toxicity graft versus host disease (GVHD) in patients with blood cancer who are undergoing donor stem cell transplant. Tacrolimus and anti-thymocyte globulin may reduce the risk of the recipient's body rejecting the transplant by suppressing the recipient's immune system. Giving bortezomib after the transplant may help prevent GVHD by stopping the donor's cells from attacking the recipient. Giving tacrolimus, bortezomib, and anti-thymocyte globulin may be a better way to prevent low toxicity GVHD in patients with blood cancer undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine a composite end point of alive and severe acute GVHD free at 6 months following human leukocyte antigen (HLA) matched related or unrelated donor hematopoietic peripheral blood transplant in patients with hematologic malignancies who receive the immunosuppressive combination tacrolimus, bortezomib, anti-thymocyte globulin (TBT) as GVHD prophylaxis.

II. To determine the safety of this combination in the first six months post-transplant.

SECONDARY OBJECTIVES:

I. To determine the cumulative incidence of grade III-IV aGVHD.

II. To determine incidence and severity of chronic GVHD.

III. To determine disease relapse or progression overall and disease free survival at one year.

OUTLINE:

Patients receive tacrolimus intravenously (IV) on day -3 through day 180. Patients may receive tacrolimus orally (PO) later at the doctor's discretion. Patients receive anti-thymocyte globulin IV on days -3, -2, and -1 and bortezomib IV on day 0 and day 3. Patients undergo allogeneic bone marrow transplant on day 0.

After completion of study treatment, patients are followed up for 6 months and then periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute leukemia, chronic myelogenous leukemia, myeloproliferative disorder and myelodysplasia with no circulating blasts and with less than 5% blasts in the bone marrow within 4 weeks of the start of transplant conditioning regimen
* Patients with chronic lymphocytic leukemia/small lymphocytic lymphoma; follicular, marginal zone, diffuse large B-cell or mantle cell lymphoma with chemo-sensitive disease at time of transplant
* Patients must have a related or unrelated peripheral blood stem cell donor; sibling donor must be a 6/6 match for human leukocyte antigen (HLA)-A and -B at intermediate (or higher) resolution, and -DRB1 at high resolution using deoxyribonucleic acid (DNA)-based typing, and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation; unrelated donor must be 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing; unrelated donor must be willing to donate peripheral blood stem cells and be medically eligible to donate stem cells according to National Marrow Donor Program (NMDP) criteria
* Cardiac function: ejection fraction > 40%
* Estimated creatinine clearance greater than 50 mL/minute (using the Cockcroft-Gault formula and actual body weight)
* Pulmonary function: carbon monoxide diffusing capability test (DLCO) ≥ 40% (adjusted for hemoglobin) and forced expiratory volume in 1 second (FEV1) ≥ 50%
* Total bilirubin < 1.5 x the upper limit of normal; patients who have been diagnosed with Gilbert's disease are allowed to exceed the defined bilirubin value of 1.5 x the upper limit of normal
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 2.5 x the upper normal limit
* Female subjects (unless postmenopausal for at least 1 year before the screening visit, or surgically sterilized), agree to practice two effective methods of contraception or agree to completely abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant
* Male subjects (even if surgically sterilized), of partners of women of childbearing potential must agree to practice effective barrier contraception or abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant
* Signed informed consent

Exclusion Criteria:

* Prior allogeneic transplant
* Karnofsky performance score < 70%
* Active central nervous system (CNS) involvement by malignant cells
* Patients with uncontrolled bacterial, viral, or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment
* Patients with transformed lymphoma (e.g., Richter's transformation arising in follicular lymphoma or chronic lymphocytic leukemia)
* Patients seropositive for the human immunodeficiency virus (HIV)
* Patient with active hepatitis B or C
* Patients with hypersensitivity to bortezomib, boron, or mannitol
* Patients with > grade 2 sensory peripheral neuropathy
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiography (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Female patients who are lactating or pregnant
* Patients with a serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Patients with prior malignancies, except resected basal cell carcinoma or treated cervical carcinoma in situ; cancer treated with curative intent > 5 years previously will be allowed; cancer treated with curative intent < 5 years previously will not be allowed unless approved by the protocol officer or one of the protocol chairs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Al-Kadhimi, MD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 9/9/2016 to 7/11/2017 at Winship Cancer Institute of Emory University.
Period: Overall Study
Arm/Group | Tacrolimus, Bortezomib, Thymoglobulin
Started | 5
Completed | 0
Not Completed | 5
Not completed — Trial was closed early | 5

BASELINE CHARACTERISTICS:
Arm/Group | Tacrolimus, Bortezomib, Thymoglobulin
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Serious Adverse Events and Adverse Events Related to This Immunosuppressive Regimen
Description: An adverse event (AE) is defined as any untoward medical experience or change of an existing condition that occurs during or after treatment. All AEs occurring during this study, whether observed by the physician, nurse, or reported by the patient, will be graded per NCI CTCAE version 4.0 and recorded on protocol-specific case report forms. A serious adverse event (SAE) is defined as any expected or unexpected adverse event (AE, generally equivalent to CTCAE grades 3, 4 or 5) that results in any of the following outcomes:
  * Death
  * Life-threatening event
  * In-patient hospitalization (not required as part of the treatment) or prolongation of existing hospitalization
  * Persistent or significant disability/incapacity
  * Congenital anomaly/birth defect
  * Cancer
  * Overdose
Time Frame: Up to 6 months post-transplant
Measure: Number; unit: events
Arm/Group | Tacrolimus, Bortezomib, Thymoglobulin
Number analyzed (Participants) | 5
events | 9

2. Primary Outcome: Number of Patients Alive and Free of Severe Acute GVHD Following HLA Matched Related or Unrelated Donor Hematopoietic Peripheral Blood Transplant
Description: Will use patient counts for the number of patients alive and free of severe acute graft versus host disease (GVHD) following human leukocyte antigen (HLA) matched related or unrelated donor hematopoietic peripheral blood transplant.
Time Frame: At 6 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus, Bortezomib, Thymoglobulin
Number analyzed (Participants) | 5
Participants | 1

3. Secondary Outcome: Cumulative Incidence of Grade III-IV aGVHD
Description: Will be summarized as percentage and 95% confidence level will be also constructed.
Time Frame: Up to 2 years post-transplant
Population: Data were not collected because trial closed early.
Arm/Group | Tacrolimus, Bortezomib, Thymoglobulin
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Chronic GVHD
Description: Will be summarized as percentage and 95% confidence level will be also constructed.
Time Frame: Up to 2 years post-transplant
Population: Data were not collected because trial closed early.
Arm/Group | Tacrolimus, Bortezomib, Thymoglobulin
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Will be analyzed with Kaplan Meier method and Logrank test.
Time Frame: At 1 year post-transplant
Population: Data were not collected because trial closed early.
Arm/Group | Tacrolimus, Bortezomib, Thymoglobulin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 180 days post-transplant.
Arm/Group | Tacrolimus, Bortezomib, Thymoglobulin
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus, Bortezomib, Thymoglobulin (N=5)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Device related infection (Infections and infestations) | 1
Confusion (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
After monitoring early toxicity and hyperacute severe acute graft versus host disease in 4/5 patients, it was decided to close this protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02877082/Prot_SAP_000.pdf